CLINICAL TRIAL: NCT02745743
Title: An Open-label, Multicenter Phase I Study to Characterize the Safety, Tolerability, Preliminary Anti-tumor Activity, Pharmacokinetics and Maximum Tolerated Dose of BAY1251152 in Patients With Advanced Hematological Malignancies
Brief Title: Phase I Trial of BAY1251152 for Advanced Blood Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18117; 2015-005122-18 (EudraCT Number)
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Hematologic Neoplasms
Keywords: Phase 1; Dose escalation; Dose expansion; Positive transcription elongation factor b inhibitor; Cyclin-dependent kinase 9 inhibitor
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Biomarker-enriched advanced hematological neoplasms
  Interventions: Drug: BAY1251152
- Arm 2 (Experimental): Other selected advanced hematological neoplasms
  Interventions: Drug: BAY1251152

INTERVENTIONS:
Drug: BAY1251152 — Weekly infusion of BAY1251152 in 21-day cycles.

SUMMARY:
The purpose of this study is to identify the most appropriate dose that can be safely administered and that can have an effect on blood cancer cells. Once that safe dose is identified, additional patients will be asked to join the study to further evaluate the safety and effectiveness of the study drug. The study will also investigate the pharmacokinetics (study of what the body does to the drug), as well as pharmacodynamics (study of what the drug does to the body), which may provide information about the effects of BAY 1251152. The study will also measure some biological markers (markers of biological activity in your body) that can be used to predict the response and safety of the proposed treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 and Life expectancy of at least 12 weeks
* Patients are able and willing to provide bone marrow biopsies/aspirates as requested by the protocol
* Patients with confirmed advanced hematological malignancies
* Negative serum pregnancy test
* Women and men of reproductive potential must agree to use highly effective contraception when sexually active.
* Ability to understand and the willingness to sign a written informed consent.
* Patients must have adequate coagulation (international normalized ratio (INR) or prothrombin time (PT), partial thromboplastin time (PTT) ≤1.5 times ULN)
* Adequate liver function (total bilirubin ≤ 1.5 times the ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN

Exclusion Criteria:

* Presence of active/uncontrolled central nervous system involvement
* History of clinically significant cardiac disease; uncontrolled hypertension
* Left ventricular ejection fraction (LVEF) < 45%
* Allogeneic stem cell transplant within 100 days before first dose of study drug
* Known history of human immunodeficiency virus (HIV) infection
* Chronic or active hepatitis B or C, requiring antiviral therapy
* Evidence of history of bleeding disorder, dialysis, or coexisting cancer that is distinct in primary site or histology from the cancer evaluated in this study
* Serious, uncontrolled infection
* Unresolved chronic toxicity > grade 1 from prior therapy
* Use of strong CYP3A4 inhibitors or strong inducers within 7 days prior to the start of study treatment and for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose(MTD) | 21 days
  To determine the MTD of BAY1251152 in subjects with advanced hematological neoplasms
Recommended Phase 2 dose (RP2D) | Up to 30 months
  To determine the RP2D of BAY1251152 based on safety, tolerability, pharmacokinetic, and pharmacodynamic data in subjects with advanced hematological neoplasms
Number of adverse events (AE) | Up to 30 months
  For assessment of the safety (ECG, vital signs, clinical significant abnormal laboratory results… etc.)and tolerability of BAY 1251152 in subjects with advanced hematological neoplasms
Pharmacokinetics (PK) is determined by maximum concentration (Cmax) | 21 days
Pharmacokinetics (PK) is determined by Area Under concentration versus time Curve (AUC) | 21 days

SECONDARY OUTCOMES:
Response assessment of BAY 1251152 in hematological malignancies based on the internationally accepted criteria for the specific hematological malignancy which patient is suffering from | Up to 30 months
  To assess the clinical efficacy of BAY 1251152 in subjects with advanced hematological neoplasms

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- United States (3):
  - New York, New York
  - The Bronx, New York
  - Nashville, Tennessee
- Dresden, Saxony, Germany
- Madrid, Spain
- Cardiff, United Kingdom

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/